CLINICAL TRIAL: NCT03366610
Title: A Long Term Off-treatment Follow-Up Study to Assess Clinical Outcomes in Chronic Hepatitis C Patients in China Previously Treated With Daclatasvir-Based Regimens
Brief Title: Study to Assess Clinical Outcomes in Chronic Hepatitis C Patients Previously Treated With Daclatasvir-Based Regimens
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI444-412
Record Dates: First submitted 2017-11-29; First posted 2017-12-08 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Patients Previously Treated with Daclatasvir-Based Regimens: Patients in China Previously Treated with Daclatasvir-Based Regimens
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Non-interventional

SUMMARY:
The purpose of this study is to assess long-term outcomes in subjects previously treated with daclatasvir-based therapy for chronic Hepatitis-C (CHC)

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age or older at initiation of prior DCV-based therapy
* Previously treated with DCV (manufactured by BMS)-based therapy in combination with other HCV direct acting antivirals (DAAs) for at least 8 weeks
* Must enroll in this study within 12 months of end of treatment of DCV-based therapy or within 6 months of protocol availability at the clinical site for subjects treated in the AI447036 or AI447114 studies

Exclusion Criteria:

- N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 1000 subjects diagnosed with CHC in China.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of hepatic disease progression events | up to 5 years

SECONDARY OUTCOMES:
Durability of virologic response | up to 5 years
  assessed by response in subjects previously treated with DCV-based therapy who achieved sustained virologic response at 12 or 24 weeks(SVR12/24) after the end of treatment
Change in liver stiffness | baseline up to 5 years
  measured using elastography values
Number of subjects with HCV sequence variants | baseline up to 5 years
  presence of HCV sequence variants over time in subjects who failed to prior Daclatasvir(DCV)-based therapy
Distribution of HCV retreatment patterns | baseline up to 5 years
  distribution of HCV retreatment patterns including number of subjects receiving retreatment, retreatment regimen, retreatment duration and retreatment results

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Beijing, Beijing Municipality, China

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm